CLINICAL TRIAL: NCT00598793
Title: Biphasic Insulin Aspart 70/30 + Metformin Compared to Insulin Glargine + Metformin in Type 2 Diabetes Failing OAD Therapy
Brief Title: Biphasic Insulin Aspart 30 in Type 2 Diabetes Failing OAD Therapy
Acronym: INITIATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-2163
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Insulin Glargine; Metformin; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: biphasic insulin aspart
Drug: insulin glargine
Drug: metformin
Drug: pioglitazone

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to compare biphasic insulin aspart 30 plus metformin in a standard injection regimen to a standard dosing of insulin glargine plus metformin on blood glucose control in subjects with type 2 diabetes who are insulin naive and failing OAD therapy.

ELIGIBILITY:
Inclusion Criteria:

* Insulin naive Type 2 diabetes
* Currently treated with OADs alone or combined with other treatment for at least 3 months
* BMI below 40 kg/m2 and body weight below 125 kg
* HbA1c greater than or equal to 8%

Exclusion Criteria:

* Inability to tolerate metformin or contradictions to its use
* Pregnant, breastfeeding or intention of becoming pregnant
* Allergy to any of the trial products
* Inability or unwillingness to perform SMBG

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2002-11; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 28 weeks of treatment

SECONDARY OUTCOMES:
Postprandial glucose by 8-point SMBG
Number of subjects achieving HbA1c below 7%
Number of hypoglycemic episodes and adverse events
Weight change
Insulin dose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (23):
- United States (23):
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Melbourne, Florida
  - Novo Nordisk Investigational Site, West Palm Beach, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Marietta, Georgia
  - Novo Nordisk Investigational Site, Idaho Falls, Idaho
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Buffalo, New York
  - Novo Nordisk Investigational Site, Asheville, North Carolina
  - Novo Nordisk Investigational Site, Canton, Ohio
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Medford, Oregon
  - Novo Nordisk Investigational Site, Hershey, Pennsylvania
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Midland, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Warrenton, Virginia
  - Novo Nordisk Investigational Site, Renton, Washington

REFERENCES:
- [Result] Raskin P, Allen E, Hollander P, Lewin A, Gabbay RA, Hu P, Bode B, Garber A; INITIATE Study Group. Initiating insulin therapy in type 2 Diabetes: a comparison of biphasic and basal insulin analogs. Diabetes Care. 2005 Feb;28(2):260-5. doi: 10.2337/diacare.28.2.260. PMID 15677776
- [Result] Garber AJ, Ligthelm R, Christiansen JS, Liebl A. Premixed insulin treatment for type 2 diabetes: analogue or human? Diabetes Obes Metab. 2007 Sep;9(5):630-9. doi: 10.1111/j.1463-1326.2006.00654.x. PMID 17697056
- [Result] Raskin P. Initiation of insulin therapy in patients with type 2 diabetes failing oral therapy: response to Mikhail and Cope and to Janka. Diabetes Care. 2005 Nov;28(11):2811. doi: 10.2337/diacare.28.11.2811. No abstract available. PMID 16249569
- [Result] Brod M, Cobden D, Lammert M, Bushnell D, Raskin P. Examining correlates of treatment satisfaction for injectable insulin in type 2 diabetes: lessons learned from a clinical trial comparing biphasic and basal analogues. Health Qual Life Outcomes. 2007 Feb 7;5:8. doi: 10.1186/1477-7525-5-8. PMID 17286868
- [Result] Ray JA, Valentine WJ, Roze S, Nicklasson L, Cobden D, Raskin P, Garber A, Palmer AJ. Insulin therapy in type 2 diabetes patients failing oral agents: cost-effectiveness of biphasic insulin aspart 70/30 vs. insulin glargine in the US. Diabetes Obes Metab. 2007 Jan;9(1):103-13. doi: 10.1111/j.1463-1326.2006.00581.x. PMID 17199725
- [Result] Raskin PR, Hollander PA, Lewin A, Gabbay RA, Bode B, Garber AJ; INITIATE Study Group. Basal insulin or premix analogue therapy in type 2 diabetes patients. Eur J Intern Med. 2007 Jan;18(1):56-62. doi: 10.1016/j.ejim.2006.09.006. PMID 17223044
- [Result] Valentine WJ, Palmer AJ, Lammert M, Nicklasson L, Foos V, Roze S. Long-term clinical and cost outcomes of treatment with biphasic insulin aspart 30/70 versus insulin glargine in insulin naive type 2 diabetes patients: cost-effectiveness analysis in the UK setting. Curr Med Res Opin. 2005 Dec;21(12):2063-71. doi: 10.1185/030079905X74989. PMID 16368057
- [Result] Goodall G, Jendle JH, Valentine WJ, Munro V, Brandt AB, Ray JA, Roze S, Foos V, Palmer AJ. Biphasic insulin aspart 70/30 vs. insulin glargine in insulin naive type 2 diabetes patients: modelling the long-term health economic implications in a Swedish setting. Int J Clin Pract. 2008 Jun;62(6):869-76. doi: 10.1111/j.1742-1241.2008.01766.x. PMID 18479280
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com